CLINICAL TRIAL: NCT03473210
Title: The Value of Amniopatch in Pregnancies Associated With Spontaneous Preterm Premature Rupture of Fetal Membranes:A Randomized Controlled Trial
Brief Title: The Value of Amniopatch in Preterm Premature Rupture of Membranes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 34
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Preterm Premature Rupture of Membrane
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes | interventions — Anti-Bacterial Agents; Adrenal Cortex Hormones; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amniopatch group (Active Comparator): in which women were subjected to active treatment included prophylactic antibiotics and antenatal corticosteroids with an effort to seal the ruptured membranes using the amniopatch technique.
  Interventions: Drug: Antibiotics; Drug: Corticosteroid; Procedure: Amniopatch
- control group (Active Comparator): in which women were subjected to conservative management with prophylactic antibiotics and antenatal corticosteroids
  Interventions: Drug: Antibiotics; Drug: Corticosteroid

INTERVENTIONS:
Drug: Antibiotics — ampicillin 2g IV every 6hours for 48 hours, followed by erythromycin 250mg every 6hours for 5days
  Other Names: ampicillin erythromycin
Drug: Corticosteroid — dexamethasone 8mg intramuscular every 12hours for 48 hours i.e. in four divided doses
  Other Names: Dexamethasone
Procedure: Amniopatch — a total of around 60-80 mL of platelets, 100-150 mL of FFP and 100-150 mL of amnioinfusion fluid was used throughout the procedure
  Arms: Amniopatch group

SUMMARY:
A randomized controlled trial that involved 100 women diagnosed with PPROM between 24 and 34 weeks of gestational age. Participants were randomized equally into 2 groups. Group I in which amniopatch was done (an amnioinfusion of platelet concentrate followed by fresh frozen plasma in addition to the routine management used in the control group. Group II were treated with routine management including antibiotics and corticosteroids

DETAILED DESCRIPTION:
All patients were started on a regimen of hospital bed rest and received antibiotic prophylaxis consisting of ampicillin 2g IV every 6hours for 48 hours, followed by erythromycin 250mg every 6hours for 5days . Antenatal corticosteroids were given in the form of dexamethasone 8mg intramuscular every 12hours for 48 hours i.e. in four divided doses.

Fifty to two hundred ml of normal saline was infused to create an adequate pocket in which the infusion needle can be stabilized. After injection of normal saline, alternate infusions of 20 mL of platelets, normal saline (which does not contain Calcium, needed for the clotting process), and 20 mL of (FFP). The infused substances were warmed to a temperature of 37°c. Avoiding contact between the blood products prevents clotting in the lines.

During infusion, the fetal heart rate as well as the accumulation of amniotic fluid was monitored by ultrasound. Usually a total of around 60-80 mL of platelets, 100-150 mL of FFP and 100-150 mL of amnioinfusion fluid was used throughout the procedure

ELIGIBILITY:
Inclusion Criteria:

* healthy pregnant women
* gestational age of 24 to 34 weeks (calculated by the sure dates of the last menstrual period and confirmed by early 1st trimesteric ultrasound).

All women carried a normal healthy singleton fetus

Exclusion Criteria:

* established preterm labor at admission
* those with symptoms or signs suggestive of clinical chorioamnionitis.
* women with uncontrolled medical disorder e.g. severe hypertension, uncontrolled diabetes, chronic renal impairment
* women with vaginal bleeding regardless its cause.
* Pregnancies associated with major congenital fetal malformations
* placental insufficiency or anomalies
* anterior position of the placenta
* iatrogenic PPROM

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-03-11 (Actual)

PRIMARY OUTCOMES:
Amniotic fluid index | one week after the procedure
  increase in amniotic fluid index to reach above the 10th percentile for the gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Study Director — professor
Locations (1):
- Hany Hassan, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided